CLINICAL TRIAL: NCT06593054
Title: An Interventional Open-Label, Single-Dose, 4-Treatment, 4-Period Crossover Study to Evaluate the Relative Bioavailability of CTB and AVI Administered Via Various Tablets or Capsule Formulations of PF-07612577 (PF-06264006 [CTB] - PF-07338233 [AVP]) and the Effect of Food on the Bioavailability of CTB and AVI Administered Via Tablets in Healthy Adult Participants
Brief Title: To Learn How Different Forms of Study Medicine Are Taken up Into the Blood and the Effect of Food on Study Medicine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C4691003; 2023-507117-10-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-07-22; First posted 2024-09-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: ceftibuten; avibactam prodrug; relative bioavailability
MeSH Terms: interventions — Ceftibuten; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CTB-AVP Capsules, fasted (Experimental): Reference formulation of CTB-AVP in capsules, administered under fasted conditions
  Interventions: Drug: Ceftibuten; Drug: Avibactam prodrug
- CTB-AVP Tablet , fasted (Experimental): Test formulation of CTB-AVP in tablets, administered under fasted conditions
  Interventions: Drug: CTB-AVP in Tablet
- CTB-AVP Tablet , fed (Experimental): Test formulation of CTB-AVP in tablets, administered under fed conditions
  Interventions: Drug: CTB-AVP in Tablet

INTERVENTIONS:
Drug: Ceftibuten — Ceftibuten dihydrate, formulated in capsules
  Arms: CTB-AVP Capsules, fasted
Drug: Avibactam prodrug — Avibactam prodrug, formulated in capsules
  Arms: CTB-AVP Capsules, fasted
Drug: CTB-AVP in Tablet — ceftibuten and avibactam prodrug, in Tablet formulation
  Arms: CTB-AVP Tablet , fasted; CTB-AVP Tablet , fed

SUMMARY:
The purpose of this study is to learn about the study medicine CTB-AVP for the treatment of severe urinary tract infections that require hospitalization.

This study is seeking for:

* adult male and female participants who are healthy and weigh more than 50 kg.
* participants who have normal blood pressure, normal kidney and liver function
* participants willing to stay away from caffeine and other medicines for the duration of the study.

Participants will be required to stay in the study clinic for two weeks. All participants in this study will receive study medicine CTB-AVP by mouth one time each day on four different days. Study medicine will be given in capsules or tablets, on an empty stomach or will be taken with a meal. The study will look at the experiences of people receiving the study medicine. This will help determine if the study medicine is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 years or older at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and standard 12-lead electrocardiogram (ECGs), and with eGFR ≥75 mL/min (estimated using the 2021 CKD-EPI equation).
2. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Have a body-mass index (BMI) of 16 to 32 kg/m2; and a total body weight >50 kg (110 lb).
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease; including any condition affecting oral absorption or known allergy to cephalosporin group of antibiotics
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention or current use of any prohibited concomitant medications.
* Screening supine Blood Pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm Hg for participants ≥60 years old, following at least 5 minutes of supine rest
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: alanine aminotransferase (ALT), aspartate aminotransferase (AST), Bilirubin ≥1.5 x Upper Limit of Normal (ULN). Participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration [Cmax] of cis-CTB and AVI following test formulation administration in fasted or fed state | Through 48 hours in period 1, 2, 3
  Cmax is estimated based on the plasma concentrations for test and reference formulation
Dose-normalized Maximum Observed Plasma Concentration [Cmax(dn)] of cis-CTB and AVI following test/ reference formulation administration | Through 48 hours in period 1, 2, 3
  Cmax is estimated based on the plasma concentrations for test and reference formulation and then normalized by dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of cis-CTB and AVI following test formulation administration in fasted or fed state | Through 48 hours in period 1, 2, 3
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Dose-Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUClast(dn)] of cis-CTB and AVI following test/ reference formulation administration | Through 48 hours in period 1, 2, 3
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) normalized by dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of cis-CTB and AVI (if data permit) following test formulation administration in fasted or fed state | Through 48 hours in period 1, 2, 3
  AUC (inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUClast plus AUClast to infinity.
Dose-Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUCinf(dn)] of cis-CTB and AVI (if data permit) following test/ reference formulation administration | Through 48 hours in period 1, 2, 3
  AUC (inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUClast plus AUClast to infinity normalized by dose

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAE) | Time the participant provides informed consent through and including follow-up contact occurring up to 35 days after the last administration of the study intervention
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is defined as any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect. AEs include both SAEs and AEs. TEAEs are AEs that occur following the start of treatment or AEs increasing in severity during treatment
Severity of treatment-emergent adverse events (TEAEs) | Time the participant provides informed consent through and including follow-up contact occurring up to 35 days after the last administration of the study intervention
Causal relationship of treatment-emergent adverse events (TEAEs) | Time the participant provides informed consent through and including follow-up contact occurring up to 35 days after the last administration of the study intervention
Withdrawals due to treatment-emergent adverse events (TEAEs) | Time the participant provides informed consent through and including follow-up contact occurring up to 35 days after the last administration of the study intervention
Number of Participants With Laboratory Abnormalities | Time the participant provides informed consent through and including follow-up contact occurring up to 35 days after the last administration of the study intervention
  Blood samples collected for the analysis of following laboratory parameters: hematology parameters (hemoglobin, erythrocyte mean corpuscular volume, erythrocyte mean corpuscular hemoglobin, erythrocyte mean corpuscular hemoglobin concentration platelet count, leukocytes, lymphocytes, neutrophils, eosinophils, monocytes); clinical chemistry parameters (bilirubin, alanine aminotransferase [ALT], blood urea nitrogen [BUN], creatinine, potassium, bicarbonate); urine parameters: urine protein, urine hemoglobin, nitrite, leukocyte esterase and bacteria. Number of participants with any laboratory abnormalities is presented.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Time the participant provides informed consent through and including follow-up contact occurring up to 35 days after the last administration of the study intervention
  Vital signs evaluation includes: supine systolic and diastolic blood pressure (BP) and pulse rate. Baseline will be the measurement taken on Day -1 and change from baseline (CFB) will be calculated for all post-baseline timepoints, and would be reported as per Sponsor's reporting standards.
Number of Participants with Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings | Time the participant provides informed consent through and including follow-up contact occurring up to 35 days after the last administration of the study intervention
  Criteria for clinically significant changes in ECG (12-lead) are defined as: a postdose QTc interval increase by ≥60 msec from the baseline and is >450 msec; or an absolute QTc value is ≥500 msec for any scheduled ECG
Time to Cmax (Tmax) of cis-CTB, AVI and hydroxypivalic acid (HPA) | Through 48 hours in period 1, 2, 3
  Tmax = time (hours) to maximum plasma concentration (Cmax).
Terminal Elimination Half-Life (t1/2) (if data permit) of cis-CTB, AVI and HPA | Through 48 hours in period 1, 2, 3
  Elimination half-life means the time required for the plasma concentration to decline by 50% during the elimination phase- if data permit
Apparent Oral Volume of Distribution (Vz/F) (if data permit) of cis-CTB, AVI and HPA | Through 48 hours in period 1, 2, 3
  Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug-If data permit
Apparent Oral Clearance (CL/F) (if data permit) of cis-CTB, AVI and HPA | Through 48 hours in period 1, 2, 3
  Clearance of a drug was measure of the rate at which the drug was metabolized or eliminated by normal biological processes- if data permit
Dose-Normalized Maximum Observed Plasma Concentration [Cmax(dn)] of HPA | Through 48 hours in period 1, 2, 3
Dose-Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUClast(dn)] of HPA | Through 48 hours in period 1, 2, 3
Dose-Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUCinf(dn)] (if data permit)of HPA | Through 48 hours in period 1, 2, 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4691003